CLINICAL TRIAL: NCT01469728
Title: Randomized Study of Thoracoscopic Talc Pleurodesis Performed by Thoracic Epidural or General Anesthesia
Brief Title: Comparison of Thoracoscopic Talc Pleurodesis by Thoracic Epidural or General Anesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Eugenio Pompeo, Associate Professor, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 107/07; #20112 (Other: TOR VERGATA UNIVERSITY)
Record Dates: First submitted 2011-10-28; First posted 2011-11-10 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Pleural Effusion
Keywords: VATS; awake thoracic surgery; pleurodesis; talc; TEA; epidural anesthesia; Video-Assisted; Anesthesia Epidural
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Awake VATS (Experimental): Thoracoscopic talc pleurodesis performed in awake patients through sole thoracic epidural anesthesia.
  Interventions: Procedure: Awake VATS talc pleurodesis
- Non-awake VATS talc pleurodesis (Active Comparator): Thoracoscopic talc pleurodesis performed through sole general anesthesia and one-lung ventilation
  Interventions: Procedure: Non-awake VATS talc pleurodesis

INTERVENTIONS:
Procedure: Non-awake VATS talc pleurodesis — Thoracoscopic talc pleurodesis performed through sole general anesthesia and one-lung ventilation
  Arms: Non-awake VATS talc pleurodesis
Procedure: Awake VATS talc pleurodesis — Thoracoscopic talc pleurodesis performed in awake patients through sole thoracic epidural anesthesia.
  Arms: Awake VATS

SUMMARY:
Video-assisted thoracoscopic surgery (VATS) talc pleurodesis is often carried out in patients with malignant recurrent pleural effusion to relieve symptoms and prevent recurrence.

General anesthesia and one lung ventilation is the standard type of anesthesia employed for VATS although recently, thoracic epidural anesthesia (TEA) in awake spontaneously ventilating patients is being increasingly employed to perform several cardio-thoracic surgery procedures in an attempt of minimize operative risks and facilitate resumption of daily-life activity.

The investigators have reasoned that for a simple and palliative procedure such as talc pleurodesis in cancer patients is, use of general anesthesia and one-lung ventilation might be considered a potential cause of morbidity and delayed recovery. The investigators have also hypothesized TEA could be considered an optimal type of anesthesia in this setting leading to a fast recovery a reduced overall workload in medical care.

In this single-center randomized study, the investigators have comparatively assessed the impact of awake TEA versus general anesthesia and one-lung ventilation on comprehensive results of VATS talc pleurodesis.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent pleural effusion at the computed tomography occupying at least 1/3 of the hemithorax in patients with recent history of malignancy.
* Karnofsky performance status ≥ 50
* ASA score II-III
* Acceptance of the randomly assigned anesthesia protocol
* Radiologic evidence of lung re-expansion after previous drainage/thoracentesis
* Absence of blood clotting disorders (INR < 1.5)
* No contraindications to TEA
* No neurological or psychiatric disturbance contraindicating awake surgery

Exclusion Criteria:

* Patients refusal of random assignment to treatment arm
* Patients refusal or noncompliance to TEA
* Patients refusal or noncompliance to general anesthesia and one-lung ventilation
* Unfavourable anatomy for TEA
* Previous surgery of the thoracic spine
* Coagulation disorders (thromboplastin time < 80%, prothrombin time > 40 sec, platelet count < 200/nL or bleeding disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-11; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Grade of perioperative medical care (PMC). | participants are followed for the duration of hospital stay; average of 5 days
  PMC is aimed at evaluating the overall workload in medical care throughout the the entire perioperative period and until discharge. PMC was computed as a comprehensive multidimensional variable including hospitalization time and extra-routine nursing/clinical/pharmacological requirements and costs(grades 1-3).

SECONDARY OUTCOMES:
Postoperative pain | Postoperatively at 3h,12h and 24h
Perioperative changes in blood gases | Imediately before operation, at end-procedure, postoperatively at 1h and 24h
  Ratio of arterial oxygen tension to fraction of inspired oxygen (PaO2/FiO2), arterial carbon dioxide tension (PaCO2)
Perioperative changes in cardiocirculatory variables including heart rate (HR) and mean arteial pressure (MAP) | Immediately before the operation, at end-procedure, postoperatively at 1h and 24h
Postoperative changes in spirometric variables | Postoperatively at 3h,12h and 24h
  Forced expiratory volume in one second(FEV1), forced vital capacity (FVC), peak expiratory flow (PEF)
Morbidity | from day of operation to discharge; average, 5 days
Hospital stay | from day of operation to discharge; average, 5 days
Redo pleurodesis | From date of operation until the date of redo pleurodesis or assessed every 6 months or until date of death from any cause
  Need of reoperation because of recurrence of the pleural effusion
Operative mortality | from day of operation for up to 30 days postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Tor Vergata University, Rome, Italy

REFERENCES:
- [Background] Pompeo E, Tacconi F, Mineo TC. Comparative results of non-resectional lung volume reduction performed by awake or non-awake anesthesia. Eur J Cardiothorac Surg. 2011 Apr;39(4):e51-8. doi: 10.1016/j.ejcts.2010.11.071. PMID 21397783
- [Background] Pompeo E, Tacconi F, Frasca L, Mineo TC. Awake thoracoscopic bullaplasty. Eur J Cardiothorac Surg. 2011 Jun;39(6):1012-7. doi: 10.1016/j.ejcts.2010.09.029. Epub 2010 Oct 25. PMID 20980159
- [Background] Vanni G, Tacconi F, Sellitri F, Ambrogi V, Mineo TC, Pompeo E. Impact of awake videothoracoscopic surgery on postoperative lymphocyte responses. Ann Thorac Surg. 2010 Sep;90(3):973-8. doi: 10.1016/j.athoracsur.2010.04.070. PMID 20732526
- [Background] Pompeo E, Tacconi F, Mineo TC. Awake video-assisted thoracoscopic biopsy in complex anterior mediastinal masses. Thorac Surg Clin. 2010 May;20(2):225-33. doi: 10.1016/j.thorsurg.2010.01.003. PMID 20451133
- [Background] Tacconi F, Pompeo E, Sellitri F, Mineo TC. Surgical stress hormones response is reduced after awake videothoracoscopy. Interact Cardiovasc Thorac Surg. 2010 May;10(5):666-71. doi: 10.1510/icvts.2009.224139. Epub 2010 Feb 23. PMID 20179134
- [Background] Tacconi F, Pompeo E, Fabbi E, Mineo TC. Awake video-assisted pleural decortication for empyema thoracis. Eur J Cardiothorac Surg. 2010 Mar;37(3):594-601. doi: 10.1016/j.ejcts.2009.08.003. Epub 2009 Sep 16. PMID 19762250
- [Background] Pompeo E, Mineo TC. Awake operative videothoracoscopic pulmonary resections. Thorac Surg Clin. 2008 Aug;18(3):311-20. doi: 10.1016/j.thorsurg.2008.04.006. PMID 18831509
- [Background] Pompeo E, Mineo TC. Two-year improvement in multidimensional body mass index, airflow obstruction, dyspnea, and exercise capacity index after nonresectional lung volume reduction surgery in awake patients. Ann Thorac Surg. 2007 Dec;84(6):1862-9; discussion 1862-9. doi: 10.1016/j.athoracsur.2007.07.007. PMID 18036900
- [Derived] Pompeo E, Dauri M; Awake Thoracic Surgery Research Group. Is there any benefit in using awake anesthesia with thoracic epidural in thoracoscopic talc pleurodesis? J Thorac Cardiovasc Surg. 2013 Aug;146(2):495-7.e1. doi: 10.1016/j.jtcvs.2013.03.038. Epub 2013 Apr 17. No abstract available. PMID 23601750